CLINICAL TRIAL: NCT06116344
Title: Improving Prostate Lesion Classification and Diagnostic Accuracy Using Machine Learning: A Comprehensive Evaluation and Development of a PI-RADS 3 Classifier
Brief Title: Improving Prostate Lesion Classification and Development of a PI-RADS 3 Classifier
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Dr. Panagiota Manava, Dr. med. Panagiota Manava, MD, senior physician, Paracelsus Medical University
Other Study IDs: AI_Prostate_1_KNN
Record Dates: First submitted 2023-08-24; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; artificial intelligence
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental: experimental: patients with a condition
- control group: control group: patients without condition

SUMMARY:
The investigators propose an AI methodology combining machine learning, histological results and expert image interpretation for the development of a PI-RADS 3 classifier.

DETAILED DESCRIPTION:
Prostate cancer is the most common carcinoma in male patients in Western industrialized countries. Multiparametric prostate MRI (mpMRI) can select patients who may be potential candidates for biopsy. In this study, the investigators present a comprehensive methodology that evaluates a multitude of AI algorithms and assesses their performance on a large and high-quality dataset, aiming to generate an efficient model and develop a PI-RADS 3 classifier. By combining the power of machine learning with the information provided by mpMRI, histopathological results as well as expert image interpretation, the investigators attempt to improve the diagnostic accuracy, which in the future my lead to more informed clinical decisions and reduce unnecessary biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Only patients with a clinical indication for mp prostate MRI will be included in this prospective study.
2. No allergies to GBCA

Exclusion Criteria:

1. Contraindications for MRI

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study population will be patients of a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Normalized Quantitative Signal - Intensity - Measurements with Region of Interest drawn in specific T2-weighted axial MRI Images | through study completion, an average of 3 years
  Regions of interest for quantitative signal intensity measurements will be drawn in various prostate lesions, the size of the region of interest will depend on the target structure. Image analysis will be performed on a PACS workstation. Signal intensity will be measured and normalized, therefore no units needed.
Quantitative Signal - Intensity - Measurements with Region of Interest in specific in Apparent diffusion coefficient (ADC) axial MRI Images | through study completion, an average of 3 years
  Regions of interest for signal intensity measurements will be drawn in various prostate lesions, the size of the region of interest will depend on the target structure. Signal intensity will be measured and normalized in mm2/s
Quantitative Signal - Intensity - Measurements with Region of Interest in specific in high b-value (800, 1500, 4000) axial MRI Images | through study completion, an average of 3 years
  Regions of interest for signal intensity measurements will be drawn in various prostate lesions, the size of the region of interest will depend on the target structure. Signal intensity will be measured and normalized in mm2/s
Signal - Intensity - Measurements with Region of Interest in specific dynamic contrast enhanced (DCE) MRI Images | through study completion, an average of 3 years
  Regions of interest for signal intensity measurements will be drawn in various prostate lesions, the size of the region of interest will depend on the target structure. Signal intensity will be measured and normalized. Image analysis will be performed on a PACS workstation. The original Time inteisity curves are transformed in relative enhancement curves. Thus, they are normalized with respect to first point in time and represent the percentage increase compared to the time before contrast arrival, no units needed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Lell, Prof. Dr. med., Study Director — Department of Radiology and Nuclear Medicine, Klinikum Nuernberg, Paracelsus Medical University, Germany
Locations (1):
- Department of Radiology and Nuclear Medicine, Klinikum Nuernberg, Paracelsus Medical University, Germany, Nuremberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566
- [Result] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Result] Morash C. What do you do with PI-RADS-3? Can Urol Assoc J. 2021 Apr;15(4):122. doi: 10.5489/cuaj.7262. No abstract available. PMID 33830009